CLINICAL TRIAL: NCT06563752
Title: Exploring the Effectiveness of Digital Anti-stigma Therapy on Illness Perception and Perceived Stigma in Patients With Schizophrenia and Their Primary Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1130113-01
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (Placebo Comparator): Before discharge, provide routine discharge preparation instructions and offer a disease education booklet with relevant health information. Follow up with two phone calls after discharge, on the 7th and 30th days.
  Interventions: Other: routine care
- Experimental (Experimental): The experimental group, referred to as the Dyad, involved both the caregiver and the patient wearing 3D glasses to watch educational VR content. The VR content included the following topics:
  1. Understanding psychiatric symptoms, including symptoms, disease course, treatment, and prognosis.
  2. Knowledge of medications and their relationship to symptom stability, as well as how to manage side effects.
  3. Schizophrenia as a chronic illness, drawing comparisons to other chronic diseases.
  4. Signs of disease relapse.
  5. How to manage persistent psychotic symptoms of schizophrenia, such as delusions, hallucinations, paranoia, and negative symptoms.
  6. How to interact and communicate with the patient.
  7. Coping with stress, stress management, and suicide prevention.
  8. Available resources.
  Interventions: Other: Participants will use 3D glasses to view VR educational information

INTERVENTIONS:
Other: Participants will use 3D glasses to view VR educational information — Participants will use 3D glasses to view VR educational information, which includes:
  1. Understanding of psychiatric symptoms, including symptoms, disease course, treatment, and prognosis.
  2. Knowledge about medications, their relationship with symptom stabilization, and handling of side effects.
  3. Schizophrenia as a chronic illness, with analogies to other chronic diseases.
  4. Signs of disease relapse.
  5. How to manage ongoing psychiatric symptoms of schizophrenia, including delusions, hallucinations, paranoia, and negative symptoms.
  6. Strategies for interacting and communicating with patients.
  7. Stress management and adjustment, as well as suicide prevention.
  8. Available resources.
  Arms: Experimental
Other: routine care — Before discharge, provide routine discharge preparation instructions and offer a disease education booklet with relevant health information. Follow up with two phone calls after discharge, on the 7th and 30th days.
  Arms: Routine care

SUMMARY:
This study aims to investigate the relationship between illness insight, self-stigma in patients with schizophrenia, and the awareness and associated stigma experienced by their families, as well as the predictors of these factors. The study will use information technology strategies for educational purposes, specifically employing 3D glasses for delivering this education. The goal is to develop a disease adaptation program that involves both patients and their families, helping to enhance disease awareness and improve stigma experiences.

DETAILED DESCRIPTION:
* Background:** Research has confirmed that family members of patients with schizophrenia often lack awareness of the illness and are affected by stigma, leading them to be reluctant to seek help. This reluctance impacts patients' medication adherence, increases the severity of the illness, and results in recurrent episodes and deteriorating social functioning. In Chinese societies, where maintaining face is important, the caregiving burden on families and associated stigma are even more pronounced. In Taiwan, there is a lack of interventions using virtual reality for family members.
* Objective:** To evaluate the effectiveness of a digital anti-stigma therapy in improving illness awareness and reducing associated stigma among patients with schizophrenia and their family members.
* Methods:** This pioneering study employs a randomized controlled trial design, involving 180 patients with schizophrenia and their family members from psychiatric medical institutions in northern Taiwan. Participants are randomly assigned to two groups: one receiving standard care and the other receiving standard care plus VR video intervention. Research tools include questionnaires on illness awareness (family and patient versions), internalized stigma scales, and family-associated internalized stigma scales. Data collection occurs at baseline, immediately post-intervention, and three months later. The t-test and χ2 test are used to assess group homogeneity, and generalized estimating equations are applied to explore the effectiveness of the intervention after controlling for basic attributes.
* Expected Results/Clinical Application:** The experimental group is anticipated to show significantly greater improvement in outcome measures compared to the control group. Implementing this intervention clinically could enhance family members' awareness of the illness and improve their experience of stigma, thereby supporting patients in adapting to their illness and stabilizing their community living.

ELIGIBILITY:
Inclusion Criteria:

Patient group

1. Age ≥ 18 years;
2. Patients who meet the DSM-5 criteria for schizophrenia or the ICD-10 diagnosis code F20, including those who are expected to be discharged from a psychiatric ward within two weeks or are outpatients;
3. Have family members involved in caregiving (i.e., relatives who assist with daily needs, supervise medication, help with medical visits, and maintain contact with hospital staff during hospitalization, including non-blood-related cohabitants);
4. Are literate, able to independently read and complete questionnaires, can operate basic tablet or smartphone functions after instruction, and are willing to participate in this study.

Family group

1. Age ≥ 18 years;
2. Family members providing care for psychiatric outpatients or inpatients diagnosed with schizophrenia (i.e., relatives who assist with daily needs, supervise medication, help with medical visits, and maintain contact with hospital staff during hospitalization, including non-blood-related cohabitants);
3. Literate, able to independently read and complete questionnaires, can operate basic tablet or smartphone functions after instruction, and are willing to participate.

Exclusion Criteria:

Patient group

(1) Patients with co-occurring personality disorders, substance or alcohol addiction, or organic brain damage; (2) Individuals living alone without close family contact; (3) Patients who will reside in a rehabilitation facility after discharge. Family group

1. Individuals with mental disorders, who are illiterate, or unable to independently read and complete questionnaires.
2. Family members who cannot use smartphones or do not have access to smart technology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  This scale primarily assesses the severity of psychiatric disorders and was originally developed by Kay et al. (1987). It includes three dimensions: positive symptoms, negative symptoms, and general psychopathology, with a total of 30 items.
The Schedule for the Assessment of Insight | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  This is a semi-structured interview questionnaire developed by David (1990), primarily used to assess illness insight and perceptions of the illness in psychiatric disorders. It includes three aspects: illness awareness, the importance of treatment, and disease recognition, with a total of 7 items.
Internalized Stigma of Mental Illness | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  This scale primarily measures the subjective self-stigma experienced by individuals with mental illness and was developed in collaboration with patients. It includes 29 items across five dimensions: alienation, stereotype endorsement, perceived discrimination, social withdrawal, and anti-stigma coping ability.
Medication Adherence Rating Scale | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  This self-report scale assesses patients' medication attitudes and adherence behaviors over the past week. It consists of 10 true/false questions, with scores ranging from 1 to 7 indicating poor adherence and 8 to 10 indicating good adherence.
Drug Attitude Inventory-10 | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  This is a self-report scale primarily used to assess patients' attitudes towards medication.
Illness Perception Questionnaire-Revised Version for Families of Patients with Schizophrenia | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  This is a survey questionnaire designed to assess illness awareness among the family members of individuals with schizophrenia. It includes 38 items across 7 dimensions, evaluating participants' knowledge about schizophrenia and its management, causes, prevalence, prognosis, and treatment.
Affiliate Stigma Scale | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  The primary purpose is to assess the caregiver's perception of internalized stigma. The scale consists of 22 items, covering three aspects: cognition, emotion, and behavior.
Caregiver Burden Scale | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  The main purpose is to assess the burden level of caregivers of psychiatric patients. The scale contains 18 questions, measuring the actual problems and feelings that arise from caregiving. The scale includes five subdimensions.
World Health Organisation- Five Well-Being Index | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  To assess the perception of Well-Being over the past two weeks.
Multidimensional Scale of Perceived Social Support | The assessment will be conducted three times: before the intervention, immediately after the intervention, and three months after the intervention.
  To assess social support from different sources. The scale consists of 12 items across three dimensions: family, friends, and significant others.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No